## Valproic Acid for Treatment of Hyperactive or Mixed Delirium in ICU

Study Protocol NCT02343575

Document Date: March 12, 2014

## Medication adjustment protocol:

## Adjustments can take place every 24 hours according to the below schedule:

If study physician decides based on the below criteria that medications need to change, they notify RA/pharmacy

| | Placebo arm | VPA arm |
|---|---|---|
| 1. start | <ul> <li>Placebo PO BID</li> <li>Rescue: HAL IV 1-5 mg</li> <li>Q4hr PRN</li> </ul> | <ul> <li>VPA PO 500 mg BID</li> <li>Rescue: HAL IV 1-5 mg</li> <li>Q4hr PRN</li> </ul> |
| 2. If ICDCS = or > 4, RASS = or > 1 and patient cont to meet criteria for hyperactive/mixed delirium, consider increasing meds according to protocol | <ul> <li>Placebo PO BID</li> <li>Rescue: HAL IV 1-5 mg</li> <li>Q4hr PRN</li> </ul> | <ul> <li>VPA 500 mg PO q am, 1000 mg PO QHS</li> <li>Rescue: HAL IV 1-5 mg Q4hr PRN</li> </ul> |
| 3. If need to increase | <ul> <li>Placebo PO BID</li> <li>Rescue: HAL IV 1-5 mg</li> <li>Q4hr PRN</li> </ul> | <ul> <li>VPA 500 mg PO q am, 1500 mg PO QHS</li> <li>Rescue: HAL IV 1-5 mg Q4hr PRN</li> </ul> |
| 4. If need to increase | <ul> <li>Placebo PO BID</li> <li>Rescue: HAL IV 1-5 mg</li> <li>Q4hr PRN</li> </ul> | <ul> <li>VPA 500 mg PO Q am, 2000 mg PO QHS</li> <li>Rescue: HAL IV 1-5 mg Q4hr PRN</li> </ul> |

- Blinded physician evaluates patient daily: clinical exam, ICDSC, DSM V criteria for delirium,
   EPS, primitive reflexes
- Research Assistant daily collects CBC (esp platelets), CMP (esp LFTs), INR, QTc, EPS side effects
- If QTC increases by 20% from initiation of medication or equals 500 or above, LFTs increase
  (ALT > 150, AST> 80) or platelets decrease by 30% or are below 150, research assistant
  consults with affiliated physician (#2). Physician #2 carefully examines situation and decides
  whether any of these changes can be due to study medication.
  - $\circ$  If No  $\rightarrow$  note is taken, study continues as designed, no unblinding necessary.
  - If Yes →study physician #1 is informed and unblinded and the best clinical decision for the patient is taken
- Patients will be in the study for total of 7 days or until resolution of delirium (ICDSC < 4 plus 24 hours), whichever is shorter time. If patients need continued treatment after the study resolution, they will be followed by the regular psychiatry consult team.</li>